CLINICAL TRIAL: NCT06002334
Title: Relationship Between Nutritional State and Respiratory Muscle Weakness in Adult Patients With Bronchietasis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Galal Salih, demonstrator, Assiut University
Other Study IDs: muscle weaknessinbroncheactsis
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To establish a relationship between malnutrion and respiratory muscle dysfunction in patients with bronchectasis

DETAILED DESCRIPTION:
Many different and prevalent chronic respiratory disorders, such as chronic obstructive pulmonary disease (COPD), cystic fibrosis (CF), non-CF bronchiectasis, idiopathic pulmonary fibrosis (IPF) and lung cancer, not only target the lungs but are often associated with systemic manifestations (1-5). The latter can be magnified by the concomitant presence of aging, comorbidities or unhealthy lifestyle habits. Nutritional abnormalities stand out amongst the systemic manifestations present in chronic respiratory conditions. When these nutritional abnormalities become very severe, with marked weight and muscle mass loss, they constitute a complex metabolic syndrome, known as cachexia. However, it should be kept in mind that the earliest stages of nutritional abnormalities do not necessarily involve evident body weight loss. Diagnosis and stratification of patients with impaired nutritional status is important to decide the appropriate therapeutic approach. In fact, it has been clearly demonstrated that therapeutic interventions, even with only moderate increases in body weight or lean mass, can improve the prognosis of respiratory patients with nutritional abnormalities (6). Therefore, medical professionals should be able to detect these deficiencies early.

One of the most important clinical consequences of nutritional deficiencies in patients with chronic respiratory disorders is the loss of muscle mass and functional impairment (2,4,9). However, nutritional deficiencies not only affect muscle mass and function, but can also have a negative impact on bone and fat tissues, reaching a state of severe cachexia in the more advanced situations. Moreover, malnutrition also targets patient's immunocompetence, facilitating infections and exacerbations, which reciprocally will contribute to worsen nutritional status.

Muscle dysfunction is defined by the loss of strength (i.e., the ability to develop a maximal effort and/or endurance (i.e., the ability to maintain a submaximal effort through time) (10,11). This functional impairment can be relatively stable (this is known as 'muscle weakness') or temporary (denominated 'fatigue', which is reversible with rest) (10,11). Muscle dysfunction can involve peripheral (limb) as well as respiratory muscles, and can appear in acute or chronic respiratory diseases due to different causes. However, the loss of muscle mass is probably the main one, at least for limb muscles, having deleterious consequences on patients' prognosis (12,13). The term 'loss of muscle mass' is generally used to express a decrease in global muscle proportion or weight, but at a cellular level it actually indicates the loss of fibers or more frequently, a reduction in their size. The loss of muscle mass is mainly because of a decrease in muscle contractile protein content through different mechanisms, including the activation of the ubiquitin-proteasome system, autophagy and apoptosis (14). Global muscle mass and fiber size are the main factors contributing to muscle strength, although other components such as fiber type proportions and muscle length also play a relevant role (12). Therefore, a loss in either muscle mass or fiber atrophy will involve a decrease in contractile strength. On the other hand, endurance depends mostly on the muscle aerobic capacity, which in turn is a subrogate of the percentage of fibers with a predominant aerobic metabolism ('slow-twitch' fibers), capillary and mitochondrial density, and the capacity of oxidative enzymes on metabolic pathways (12).

The presence of limb muscle dysfunction can even limit normal walking, leading to a reduction of patient daily activities and social life, with a strong negative impact on prognosis, quality of life, and utilization of social and health resources (3,7,8,15-18). Respiratory muscle dysfunction in turn is associated with increased dyspnea (10,11,19), a worse ventilatory response to both exercise and exacerbations (19-21), and can even lead to severe respiratory failure, as well as weaning difficulties in patients submitted to mechanical ventilation (22,23).

Bronchiectasis, defined as the abnormal and irreversible dilation of the bronchi, are frequently observed even in general population, especially since the wide use of the high-resolution computed tomography (122). Although bronchiectasis can be the result of different processes, they are currently classified in those linked to CF and those that are independent of such a genetic alteration (non-CF), being the latter much more prevalent (123-125). Moreover, the above-mentioned advances in image techniques have allowed for the identification of a variable number of COPD patients who also have bronchiectasis to a greater or lesser extent (1). Although the most common clinical presentation of non-CF bronchiectasis is the presence of daily cough with abundant sputum and repeated infections (123,124), nutritional abnormalities are also frequent (2). Since many of the deleterious factors present in COPD are also present in non-CF bronchiectasis (local and systemic inflammation, exacerbations, ventilatory limitation, deconditioning, etc.) (126,127), it could be speculated that muscle dysfunction would also be frequent in this case. However, the actual prevalence of this disorder in non-CF bronchiectasis remains unclear. Respiratory muscle dysfunction has only been occasionally described in this lung disease (2,126,128,129) and, so far little attention has been given to the eventual presence of limb muscle malfunctioning. In fact, only isolated reports suggest that this latter abnormality is common in non-CF bronchiectasis (130,131) and exercise tolerance can also be reduced (126).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders who have bronchiectasis based on imaging

Exclusion Criteria:

Patients less than 18 years old Patients with neuromuscular disorders, muscle dystrophies or other causes of muscle weakness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient with bronchectasis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-04-23 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
To establish a relationship between malnutrion and respiratory muscle dysfunction in patients with bronchectasis | 1 year
  To establish a relationship between malnutrion and respiratory muscle dysfunction in patients with bronchectasis

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Assiut University, Asyut, Egypt